CLINICAL TRIAL: NCT04844515
Title: The ESPERES Prospective Cohort of Healthcare Workers in France: Study on COVID-19 Vaccine and the COVID-19 Pandemic
Brief Title: The ESPERES Prospective Cohort of Healthcare Workers in France: Study on COVID-19 Vaccine and the COVID-19 Pandemic (ESPERES_COVID19)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210173.1
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthcare Workers; COVID-19
Keywords: Healthcare workers; Preventive measures; Attitudes; COVID-19
MeSH Terms: conditions — COVID-19; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the first study performed within the ESPERES cohort, related to prevention against COVID-19, in particular vaccination against COVID-19 and more broadly on the COVID-19 pandemic.

ESPERES is a national prospective e-cohort study providing a resource for collecting information on healthcare workers (HCWs) currently working in France. The overall goal of ESPERES is to develop the infrastructure necessary to create and engage a community of HCWs who may be eligible for participation in future research studies. ESPERES is set up to answer research questions, in the field of prevention for HCWs, prevention for their own health, that of their relatives, their colleagues, and users of the hospital. These research questions will be carried out in the context of specific subsequent studies.

DETAILED DESCRIPTION:
Most countries face the issue of vaccine hesitancy, with sizeable fractions, or sometimes the majority, of the public opposing some vaccines. The problem is particularly acute in the case of COVID-19 vaccination: first, a high uptake of COVID-19 vaccines is necessary to reach and sustain herd immunity; second, and to the best of our knowledge, no country is currently planning on making COVID-19 vaccination mandatory, making public approval essential. Unfortunately, hesitancy towards COVID-19 vaccines is high in many countries.

Vaccine hesitancy also concerns healthcare workers (HCWs) who are at the frontline of the COVID-19 pandemic and identified as a priority target group for COVID-19 vaccines. Furthermore, HCWs can be relays of information concerning vaccination and thus play a key role as mediator in the promotion (or not) of this vaccination. However, vaccine intentions against COVID-19 are not fully known among different categories of HCWs and are likely to evolve with knowledge about the safety and efficacy of vaccines as well as the evolution of the epidemic. Consequently, it is crucial to understand the evolution of these vaccine intentions and their determinants in HCWs in order to better target interventions to promote this vaccination, in a context where scientific data are themselves evolving quickly.

The study population will be made up of HCWs. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.). ESPERES_COVID-19 will be offered to all the HCWs of the Assistance Publique - Hôpitaux de Paris (AP-HP) establishments and to other public or private health establishments (lucrative or not) in the Ile-De-France region and to establishments in other French regions, in order to diversify the contexts.

Each participant is self-included and collects his own data via a web interface. This cohort is open, meaning that eligible people can be included until the end of the study (no limited inclusion period). This cohort will start in 2021 and is scheduled for an initial duration of 24 months but may be extended as part of amendments.

Participants will be regularly asked to answer online questionnaires lasting at most 20 minutes. The frequency of these questionnaires will not exceed one questionnaire every 2 weeks (and will generally be more spaced out). During their follow-up in the cohort, participants may be asked, depending on their characteristics, to participate in studies nested in the cohort.

All data from ESPERES_COVID-19 will be gathered in a health data repository. The statistical analyses planned in the research protocol will be performed by the pharmaco-epidemiology center (CEPHEPI), under the responsibility of Dr Candice ESTELLAT and Pr Florence TUBACH. The CEPHEPI is backed by the public health department of the hospital group Pitié-Salpêtrière - Charles Foix, AP-HP.

A calculation of the sample size is not justified for this study as it aims to answer several research questions in a cohort. However, a number about 15,000 participants in ESPERES_COVID-19 are expected.

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Healthcare workers defined as individuals who currently work in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.)
* Agreeing to participate (digital consent)

Exclusion Criteria:

- No internet access

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of HCWs. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.). ESPERES_COVID-19 will be offered to all the HCWs of the Assistance Publique - Hôpitaux de Paris (AP-HP) establishments and to other public or private health establishments (lucrative or not) in the Ile-De-France region and to establishments in other French regions, in order to diversify the contexts.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-04-23 (Estimated)

PRIMARY OUTCOMES:
The COVID-19 vaccine intention with the question: "Do you intend to get vaccinated against COVID-19?" : I am already vaccinated / Yes, as soon as possible / Yes, but I prefer to wait before getting vaccinated / No, I don't think I'm gonna get vaccinated | Up to 24 months

SECONDARY OUTCOMES:
The COVID-19 vaccine intention in HCWs participants according to the characteristics of the vaccines (country of the manufacturer, technology used, number of doses, etc.) and of the HCWs | Up to 24 months
Potential individual sociocognitive factors in the acceptance of COVID-19 vaccination, based on models developed for vaccine hesitation (5C psychological antecedents of vaccination adapted for COVID-19 vaccination and HCWs). (eleven points-Likert scales) | Up to 24 months
The perceptions of participants regarding the strategies for managing the pandemic and the progress of the health crisis and the pandemic (eleven points-Likert scales) | Up to 24 months
The healthy behaviors in other contexts (especially influenza vaccination over the last years) | Up to 24 months
The methods and sources of information concerning questions relating to health: media (website, social networks, television, radio or written press), nature (mainstream, classic or alternative media), etc. | Up to 24 months
Frequency of searches for information on COVID-19 or COVID-19 vaccines | Up to 24 months
Socio-demographic and professional characteristics, lifestyles: age, gender, profession and place of practice | Up to 24 months
The percentages of participants with history of COVID-19 and risk factors for severe forms of COVID-19 (perception of being at risk for severe forms) | Up to 24 months
The impact of the epidemic on the participants in their professional and personal life (closed-ended questions) | Up to 24 months
Contextual determinants: characteristic of living (density and constitution of the household) and work (type of hospital, working hours, time and mode of travel to workplace) places | Up to 24 months
Other health behaviors related to the COVID-19 pandemic: adherence to protective measures in professionnal and personal life during the last 14 days (eleven points-Likert scale) | Up to 24 months
The self-reported COVID-19 vaccine rate (dates, number of doses, type of vaccine, satisfaction) | Up to 24 months
Incidence of SARS-COV-2 infection (date, severity, mode of diagnosis, etc.) | Up to 24 months
The attitude of HCWs participants regarding the advice they give or not to patients, relatives and colleagues regarding the vaccination against COVID-19 (closed-ended questions) | Up to 24 months
Behavioral risk factors during the last 14 days before the SARS-COV-2 infection (closed-ended questions) | Up to 24 months
Other health behaviors related to the COVID-19 pandemic: the frequency of carrying out diagnostic tests for the infection to SARS-COV-2 | Up to 24 months
The perceptions of participants in general regarding to the COVID-19 vaccination (eleven points-Likert scales) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence Tubach, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière - Charles Foix, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided